CLINICAL TRIAL: NCT05499663
Title: Leveraging Technology to Address POST-Treatment Health Outcomes of Cancer Survivors (POSTHOC-II): A Phase II Survivorship Care Plan Randomized Controlled Trial
Brief Title: Title: Leveraging Technology to Address Health Outcomes of Cancer Survivors
Acronym: POSTHOC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Charles River Analytics (Industry)
Responsible Party: Principal Investigator, Amber Kleckner, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00100473; 75N91021C00019-0-9999-1 (NIH)
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Results first posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Survivorship; Cancer; Symptoms and Signs
Keywords: mobile health; mhealth; exercise; nutrition; behavior change
MeSH Terms: conditions — Neoplasms; Signs and Symptoms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POSTHOC app (Experimental)
  Interventions: Behavioral: POSTHOC app
- Control (No Intervention)

INTERVENTIONS:
Behavioral: POSTHOC app — The POSTHOC app is a smartphone application that will deliver the Survivorship Care Plan and promote healthy lifestyle behaviors consistent with the individual's Care Plan
  Arms: POSTHOC app

SUMMARY:
At the end of cancer treatment, many patients are still dealing with symptoms of cancer and side effects of treatment. Many are also left in a surreal mental state with uncertainty regarding the future of their health. Survivorship Care Plans are plans that are provided to individuals at the completion of cancer treatment (i.e., chemotherapy, surgery, radiation). Survivorship Care Plans describe the details of a person's diagnosis and treatment, as well as provide recommendations for follow-up appointments, referrals, and healthy behaviors to accelerate recovery and prevent recurrence (e.g., diet, exercise, smoking cessation). Survivorship Care Plans are currently static documents that are provided via paper and become outdated as soon as the person's health status changes. Therefore, there is a need to digitize Survivorship Care Plans to improve the accessibility, modifiability, and longevity of the plan. In addition, with current technology, there is an opportunity for Survivorship Care Plans to be linked with mobile devices and activity trackers so that people can track health behaviors and compare them to their clinical goals, enabling people to take charge of their own health. Charles River Analytics developed an app called POSTHOC (POST-treatment Healthcare Outcomes for Cancer survivors) that digitizes the Survivorship Care Plan with goals to integrate it into the digital medical record.

Herein, phase I/II feasibility/preliminary efficacy randomized controlled trial is being conducted among 54 patients with cancer who recently completed adjuvant treatment for cancer (e.g., chemotherapy, radiotherapy, surgery) to compare 12 weeks of the POSTHOC app as part of the Survivorship Care Plan vs. the usual care Survivorship Care Plan on total symptom burden. Participants will be randomized 2:1, POSTHOC:usual care. All participants will be asked to download the POSTHOC app to assess technical compatibility and for data collection purposes (i.e., step count via Fitbit, ecological momentary assessment). All participants will have a "lite" version of the app for baseline. Upon randomization, those randomized to the POSTHOC group will be provided with their Survivorship Care Plan via the app, and will choose to focus on nutrition or exercise for the duration of the study, based on their individual plan and personal preferences. These features will also become accessible in the app. At baseline, 6 weeks, and 12 weeks, patient-reported outcomes will be evaluated including total symptom burden, diet, and physical activity. Extensive quantitative and qualitative feedback will also be collected on the usability of the app from those in the POSTHOC arm in order to improve the app for future implementation studies.

ELIGIBILITY:
Inclusion Criteria:

* Have had a cancer diagnosis (any type)
* Will soon or have recently completed treatment (within the past 12 weeks) with chemotherapy, radiotherapy, or surgery with curative intent
* Must have received, plans to receive, or open to receiving a Survivorship Care Plan (SCP) as per their provider
* Have access to a device capable of running the POSTHOC app and Fitbit app (e.g., Android or Apple smartphone) and reliable Internet access
* Be at least 18 years of age
* Be able to read and understand English, and
* Be able to provide written informed consent

Exclusion Criteria:

* Have planned surgery, radiotherapy, or surgery during the study period (hormonal and biologic therapy is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amber Kleckner, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] James S, Clingan CL, Adesanya IA, Zhu S, Francis ME, Rosenblatt PY, Molitoris JK, Deighton DC, Winder AT, Desrochers PC, McGeorge NM, Kleckner IR, Kleckner AS. Leveraging technology to address POST-Treatment Health Outcomes of Cancer Survivors (POSTHOC): A phase I/II randomized controlled trial of a survivorship care plan mobile application. J Cancer Surviv. 2025 Nov 27:10.1007/s11764-025-01946-7. doi: 10.1007/s11764-025-01946-7. Online ahead of print. PMID 41307872
- [Derived] Chung KH, Youngblood SM, Clingan CL, Deighton DC, Jump VA, Manuweera T, McGeorge NM, Renn CL, Rosenblatt PY, Winder AT, Zhu S, Kleckner IR, Kleckner AS. Digitizing Survivorship Care Plans Through the POST-Treatment Health Outcomes of Cancer Survivors (POSTHOC) Mobile App: Protocol for a Phase II Randomized Controlled Trial. JMIR Res Protoc. 2024 Sep 5;13:e59222. doi: 10.2196/59222. PMID 39235855

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completion of baseline assessments was necessary before randomization
Groups:
- Control: Usual care
Period: Overall Study
Arm/Group | POSTHOC App | Control
Started | 23 | 11
Completed | 22 | 10
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | POSTHOC App | Control | Total
Number analyzed (Participants) | 23 | 11 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (10.2) | 57.5 (13.6) | 61.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 8 | 27
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 20 | 10 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 11 | 34
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Logged Data at Least Three Times in the POSTHOC App
Description: Number of participants who logged data at least three times in the POSTHOC app
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- POSTHOC App: The POSTHOC app is a smartphone application that will deliver the Survivorship Care Plan and promote healthy lifestyle behaviors consistent with the individual's Care Plan. These participants will have access to the following features of the POSTHOC app: their individualized Survivorship Care Plan, recommendations for daily step count and a comparison of their actual (via Fitbit) vs. their goal, recommendations for daily food groups and a comparison to their actual (entered manually) to their goal, symptom logging, and Ecological Momentary Assessment
- Control: Usual care. These participants downloaded the POSTHOC app, but only had access to the Ecological Momentary Assessment feature of the app.
Arm/Group | POSTHOC App | Control
Number analyzed (Participants) | 23 | 11
Participants | 12 | 1

2. Primary Outcome: Usefulness of POSTHOC App
Description: 7-point Likert scale for usefulness flanked by 1=not at all useful and 7=extremely useful
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | POSTHOC App
Number analyzed (Participants) | 18
points | 3.4 (2.0)

3. Primary Outcome: Usefulness of POSTHOC App
Description: 7-point Likert scale for usefulness flanked by 1=not at all useful and 7=extremely useful
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | POSTHOC App
Number analyzed (Participants) | 19
points | 4.3 (2.3)

4. Primary Outcome: Likely to Recommend the POSTHOC App
Description: 7-point Likert scale flanked by 1=not at all likely to recommend to others and 7=extremely likely
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | POSTHOC App
Number analyzed (Participants) | 18
points | 4.2 (2.2)

5. Primary Outcome: Likely to Recommend the POSTHOC App
Description: 7-point Likert scale flanked by 1=not at all likely to recommend to others and 7=extremely likely
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | POSTHOC App
Number analyzed (Participants) | 19
points | 4.4 (2.3)

6. Secondary Outcome: Cumulative Symptom Burden
Description: This is a sum of severities of the core patient-reported symptoms from the MD Anderson Symptom Inventory, including fatigue, insomnia, pain, appetite loss, dyspnea (shortness of breath), cognitive problems, nausea, distress, and sensory neuropathy. The scale ranges from 0-130. A higher score indicates higher symptom burden.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | POSTHOC App | Control
Number analyzed (Participants) | 21 | 9
points | 20.0 (20.8) | 18.6 (18.3)

7. Secondary Outcome: Cumulative Symptom Burden
Description: as for outcome 6
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | POSTHOC App | Control
Number analyzed (Participants) | 21 | 9
points | 19.8 (21.4) | 26.7 (21.7)

ADVERSE EVENTS:
Time Frame: From enrollment to the end of 12 weeks
Groups:
- Before Randomization: Participants who consented to the study but then withdrew before randomization
Arm/Group | POSTHOC App | Control | Before Randomization
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/11 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/11 | 1/17
Other Adverse Events (participants affected / at risk) | 0/23 | 1/11 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | POSTHOC App (N=23) | Control (N=11) | Before Randomization (N=17)
Cancer metastasis (Nervous system disorders) | 0 | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | POSTHOC App (N=23) | Control (N=11) | Before Randomization (N=17)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
For 10 consented participants, app download was unsuccessful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT05499663/Prot_SAP_ICF_000.pdf